CLINICAL TRIAL: NCT05839912
Title: Lymph Node Excision (LNEx) for Patients With Stage III Melanoma With One Clinically Positive Node: Excision of Lymph Node Trial [EXCILYNT]
Brief Title: Excision of Lymph Node Trial (EXCILYNT) (Mel69)
Acronym: EXCILYNT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Craig L Slingluff, Jr (Other)
Responsible Party: Sponsor-Investigator, Craig L Slingluff, Jr, Principal Investigator, University of Virginia
Organization: University of Virginia (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 230011
Record Dates: First submitted 2023-04-20; First posted 2023-05-03 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Melanoma
Keywords: melanoma; surgery; lymph node excision
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1: Excision of cLN before systemic therapy (Experimental): Excision of the clinically detected metastatic lymph node before systemic therapy.
  Interventions: Procedure: Excision of clinically detected lymph node metastasis before any systemic therapy
- Cohort 2: Excision of cLN after neoadjuvant systemic therapy (Experimental): Excision of the clinically detected metastatic lymph node after systemic neoadjuvant therapy.
  Interventions: Procedure: Excision of clinically detected lymph node metastasis after neoadjuvant systemic therapy

INTERVENTIONS:
Procedure: Excision of clinically detected lymph node metastasis before any systemic therapy — Surgical intervention to remove the clinically detected lymph node metastasis after which physician choice adjuvant systemic therapy is permitted
  Arms: Cohort 1: Excision of cLN before systemic therapy
Procedure: Excision of clinically detected lymph node metastasis after neoadjuvant systemic therapy — Surgical intervention to remove the clinically detected lymph node metastasis after physician choice neo adjuvant systemic therapy. Physician choice adjuvant therapy is allowed after surgery
  Arms: Cohort 2: Excision of cLN after neoadjuvant systemic therapy

SUMMARY:
The purpose of this study is to find out if removing only the cancerous lymph node (known as a lymph node excision) is effective at preventing cancer from coming back in the same area of the lymph node excision. The study team is also trying to find out the side effects of this type of surgery and how much the surgery impacts quality of life.

In order to be eligible for this study, participants must have been diagnosed with metastatic melanoma and have one detected cancerous lymph node by imaging (CT/PET scan) or clinical examination, and are a candidate for lymph node excision.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, aged 18 years or older at enrollment
4. ECOG performance status of 0-2
5. Subjects must have histologically (or cytologically) confirmed metastatic melanoma to only one lymph node in the axilla, groin, or iliac basin that was detected clinically. A clinically positive lymph node is defined as a palpable and clinically suspicious node (based on palpation or imaging), or non-palpable lymph node that is FDG-avid or ≥ 0.95 cm on PET-CT, based on professional assessment of the radiologist, and that also is confirmed to contain metastatic melanoma on biopsy.

   a) The clinically positive lymph node may have been removed within 8 weeks prior to enrollment, and in that case may or may not have been evaluated by PET-CT; it is considered a clinically positive node if it was either identified as clinically suspicious on exam and/or on preoperative scans based on FDG-avidity and/or diameter ≥ 0.95 cm, and also confirmed histologically. The clinically positive node must be within the primary draining node basin of the primary melanoma, or the metastasis may be from an unknown primary site. A node that was removed at sentinel node biopsy will not meet this eligibility criterion. A patient will not be eligible if there is evidence of an additional clinically positive node on imaging or physical exam after excision of the first clinically positive node.
6. Subjects must be able to undergo LNEx and must not be on a clinical trial that requires TLND.

   a. Subjects may have previously had metastatic melanoma to a sentinel node in the same node basin, if complete lymph node dissection was not done, and if at least 1 year has elapsed since the prior positive sentinel node biopsy.
7. Individuals will be required to have radiological studies to rule out radiologically evident melanoma metastasis. Required studies include:

   * PET-CT scan, and
   * Head CT scan or MRI These scans may have been performed prior to resection of the primary melanoma and/or sentinel node biopsy if they showed no evidence of other metastases.

Exclusion Criteria:

1. Subjects who have had a prior complete lymph node dissection or radiation therapy of the clinically positive node basin.
2. Subjects who have, or have had, in-transit or satellite metastases from the same primary melanoma that has metastasized to the cLN that is the focus of the current study.

   a. The only exception are subjects who have had in-transit or satellite metastases without intervening recurrence within the year prior to the subject's enrollment on the study.
3. Subjects who have, or have had, one or more metastases distant to the primary draining lymph node basin. An individual with small radiologic or clinical findings of an indeterminate nature may still be eligible: examples include a new 5 mm lung nodule that is too small to characterize or an asymptomatic 12 mm bony lucency that is not classic for malignancy, where clinical care may otherwise be to follow the patient with repeat imaging rather than to treat the lesion.
4. Subjects with pre-existing lymphedema that precludes assessment of lymphedema. Pre-existing lymphedema should be discussed with the principal investigator (PI) at the treating institution or the overall study PI. Some patients with mild stable lymphedema at the time of enrollment may still be evaluable. The primary endpoint for lymphedema measurement is the circumference 10 cm proximal to ankle/wrist on the involved side vs the contralateral side. If there is a pre-existing difference, then it will be important to be able to assess for meaningful increases after surgery.
5. Subjects whose treating physician(s) plan adjuvant radiation therapy to the involved node basin, because that also would confound assessment of node basin recurrence and lymphedema.
6. Individuals for whom there is a medical contraindication or potential problem in complying with the requirements of the protocol in the opinion of the investigator.
7. Subjects with a prior or concurrent malignancy may be eligible if its natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the regimen.
8. Subjects who are receiving systemic or intratumoral therapy for this melanoma within 3 months of enrollment. They may have received prior adjuvant systemic therapy for an earlier stage of disease, but should be off that therapy for 3 months prior to enrollment.

   1. The only exception is for patients who are being treated at a participating center with neoadjuvant therapy for 1 cLN, and who otherwise meet criteria for enrollment. They should be screened and enrolled as soon as possible. The intent of this exception is to allow enrollment of patients who are being evaluated at that center before the study is open but whose LN Excision date can occur after the study is open to enrollment, or for patients who are not able to make a decision about enrollment on this study prior to starting neoadjuvant therapy. For such patients, data collected prior to starting neoadjuvant therapy should be recorded as screening data (such as imaging studies), but baseline lymphedema measurements, FACT-M and WPAI surveys, and anything else not done prior to starting neoadjuvant therapy should be performed as soon as possible, and prior to LN Excision. This exception does reduce the power to address some exploratory endpoints; so, use of this exception should be minimized as much as possible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Node basin-only recurrence | 3 years after the lymph node excision
  Number of participants with recurrence of melanoma within the node basin without concurrent or preceding distant metastatic recurrence

SECONDARY OUTCOMES:
Lymphedema | within 3 years after the lymph node excision
  Proportion of patients with lymphedema in the extremity closest to the dissected lymph node basin

CONTACTS AND LOCATIONS:
Overall Officials: Craig L Slingluff, Jr., MD, Principal Investigator — University of Virginia
Locations (7):
- United States (7):
  - Emory University, Atlanta, Georgia
  - University of Maryland, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Health System, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Cancer Center at the University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No